CLINICAL TRIAL: NCT02969096
Title: Evaluating the Safety and Efficacy of Targeted Cryoablation Therapy in the Treatment of Hepatic Carcinoma
Brief Title: Clinical Study of Targeted Cryoablation Therapy in the Treatment of Hepatic Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAA
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Liver Neoplasms
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Targeted Cryoablation Therapy (Experimental): liver cancer patients received targeted cryoablation therapy.
  Interventions: Procedure: Targeted Cryoablation Therapy

INTERVENTIONS:
Procedure: Targeted Cryoablation Therapy — A cryoprobe is inserted percutaneously under CT guidance into the targeted lesion. Patients undergo ablation using a freeze-thaw-freeze cycle lasting approximately 6-10-6 or 8-10-8 minutes, respectively.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of targeted cryoablation therapy for hepatic carcinoma.

DETAILED DESCRIPTION:
A cryoprobe is inserted percutaneously under CT guidance into the targeted lesion. Patients undergo ablation using a freeze-thaw-freeze cycle lasting approximately 10-6-10minutes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of liver cancer based on histology or the current accepted radiological measures.
* Single Tumor size ≤5.0 cm in greatest diameter, or multiple tumor number≤3 and each tumor size≤ 3cm.
* Life expectancy: Greater than 3 months.
* Patients' liver function is Child-pugh A or B.
* Ability to understand the study protocol and a willingness to sign a written informed consent document.
* Unable to receive operative surgery.

Exclusion Criteria:

* Patients with other primary tumor except liver cancer.
* History of coagulation disorders or anemia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Rate of complete tumor ablation | Up to 4 weeks post surgery

SECONDARY OUTCOMES:
Adverse Events | Up to 4 weeks post surgery

CONTACTS AND LOCATIONS:
Overall Officials: qing wu, Bachelor, Study Director — Shanghai Longhua Hospital
Locations (1):
- Shanghai Longhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided